CLINICAL TRIAL: NCT05268783
Title: Patient-reported Outcomes in Neuroendocrine Neoplasms: a Prospective Quality of Life and Quality of Care Study Within NETwerk
Acronym: Quali-NET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Quali-NET
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-02

CONDITIONS: Quality of Life
Keywords: neuroendocrine neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEN patients (Experimental): EORTC QLQ-C30, EORTC QLQ-GI.NET21 and satisfaction survey
  Interventions: Procedure: EORTC QLQ-C30; Procedure: EORTC QLQ-GI.NET21; Procedure: Satisfaction survey

INTERVENTIONS:
Procedure: EORTC QLQ-C30 — Quality of life questionnaire that has to be completed every 6 months
Procedure: EORTC QLQ-GI.NET21 — Quality of life questionnaire that has to be completed every 6 months
Procedure: Satisfaction survey — Questionnaire regarding satisfaction of care that has to be completed on Day 1.

SUMMARY:
Neuroendocrine tumors (NET) are rare tumors that require specific diagnosis and treatment. Therefore, this poses a challenge for clinical practice. Diagnosis and treatment can be optimized when physician specialists and other healthcare providers, across various hospitals, join forces to provide patients the best care. Based on this idea, a hospital network called NETwerk was set up. The following hospitals are part of this network: University Hospital Antwerp, VITAZ, AZ Monica, AZ Voorkempen, AZ Klina, Gasthuiszusters Antwerpen, Ziekenhuis Netwerk Antwerpen and AZ Rivierenland. In this NETwerk, patients with a neuroendocrine tumor or patients suspected with a neuroendocrine tumor are discussed with the specialists and treated.The aim of this study is to map the quality of life of NET patients within NETwerk in order to optimize the quality of care. Throughout the diagnosis, the treatment process and the follow-up, the patient will be asked to fill out three questionnaires (QLQ-C30, QLQ-GI.NET21 and a satisfaction survey). These questionnaires will be filled out every six months at home. Patients will be asked to complete these questionnaires over a period of five years.

ELIGIBILITY:
Inclusion Criteria:

* NEN patient
* 18 years or older
* Patient should appear in Oncobase

Exclusion Criteria:

* Patients who do not have an email address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life measurement with QLQ-C30 questionnaire | 5 years
  Quality of life measurement with QLQ-C30 questionnaire
Quality of life measurement with QLQ-GI.NET21 questionnaire | 5 years
  Quality of life measurement with QLQ-GI.NET21 questionnaire

SECONDARY OUTCOMES:
Quality of care measurement with satisfaction survey | 5 years
  Quality of care measurement with satisfaction survey

CONTACTS AND LOCATIONS:
Locations (7):
- Belgium (7):
  - AZ Klina, Brasschaat, Antwerp
  - AZ Monica, Deurne, Antwerp
  - Antwerp University Hospital, Edegem, Antwerp
  - AZ Rivierenland, Rumst, Antwerp
  - VITAZ, Sint-Niklaas, East-Flanders
  - ZNA, Antwerp
  - GZA, Antwerp

IPD SHARING:
Plan to Share IPD: No